CLINICAL TRIAL: NCT00398918
Title: Alcohol Self Administration Laboratory
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: H-25360
Record Dates: First submitted 2006-11-13; First posted 2006-11-14 (Estimated); Results first posted 2010-05-14 (Estimated); Last update posted 2017-07-14 (Actual); Status verified 2017-06

CONDITIONS: Alcoholism
MeSH Terms: conditions — Alcoholism | interventions — Zonisamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zonisamide (Experimental)
  Interventions: Drug: zonisamide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: zonisamide — zonisamide (100 mg)one time
  Other Names: zonegran
  Arms: Zonisamide
Drug: Placebo — Placebo Comparator
  Arms: Placebo

SUMMARY:
This is a pilot study in which our intent is to establish an alcohol administration laboratory in which we will be able to test the effect of the anticonvulsant medication zonisamide as compared to placebo on alcohol self administration and on cognitive functioning in non treatment seeking heavy users of alcohol. Our first goal is to establish the safety of zonisamide when used together with alcohol. Our second goal is to test the effect of an acute dose of zonisamide on alcohol consumption and show that it may reduce the consumption of alcohol. To achieve this goal we seek subjects with a history of heavy drinking to be tested on the self-administration procedures described below in two sessions with either zonisamide or placebo. These procedures will involve first, the administration of a challenge dose of ethanol to evaluate the effect of alcohol on performance on neuropsychological tests. This initial challenge will be followed by a period of alcohol self-administration in which the research subject can choose to select either ethanol or another reinforcer, money.

DETAILED DESCRIPTION:
In preclinical studies three novel anticonvulsants have been studied. The administration of tiagabine did not decrease ethanol consumption in rodents (Schmitt et al., 2002; Rimondini et al., 2002). In a study with alcohol preferring mice topiramate reduced alcohol consumption in a two bottle choice prolonged access model of drinking (Gabriel and Cunningham, 2005). In a study done at our laboratory both topiramate and zonisamide were found to have similar effects on reducing the consumption of ethanol in Wistar rat (Knapp et al., 2004). More recently we found that zonisamide administration decreased alcohol consumption in a limited access model in the C57BL/B6 mouse. These results suggest that zonisamide might be useful as a medication for the treatment of alcohol dependence.

Topiramate and zonisamide have some structural similarities with a sulfamate or methane-sulfonamide containing chain respectively attached to cyclic structure. These structural similarities may explain some of their pharmacological similarities including blockade of voltage sensitive sodium channels and low potency inhibition of carbonic anhydrase (Taverna et al., 1999; Dodgson et al., 2000; Schaf et al., 1987; Masudaet al., 1993). Both topiramate and zonisamide promote weight loss (McElroy et al., 2003; McElroy et al., 2004; Gadde et al., 2003). This effect may be a result of neuromodulation of the regulation of alcohol and food shared by these drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Non treatment seeking subjects ages 21-55 must indicate no treatment for alcohol dependence in the preceding 6 months.
2. Male subjects must drink no more than 40 standard drinks; female subjects no more than 35 standard drinks a week as determined by the TLFB
3. Subjects must be able to provide IC
4. BAC must be 0.000 at the time of consent
5. Female subjects of a child bearing potential must use an acceptable method of contraception which includes a barrier and spermicide, levonorgestrel implant, medroxyprogesterone, intrauterine progesterone contraceptive system or complete abstinence or surgical sterilization. Women who are using oral contraceptives must agree to an additional barrier method.

Exclusion Criteria:

1. Subject meeting DSM-IV-TR criteria for axis I diagnosis that require pharmacological treatment.
2. Subject meeting substance dependence criteria for any substance other than alcohol or nicotine .
3. Positive urine toxicology screen for opioids, cocaine, amphetamines, PCP, THC (may repeat THC if positive).
4. History of severe alcohol withdrawals.
5. Any medical or psychological condition that in the opinion of the investigator will preclude safe participation in the trial. These include a history of kidney stones in the past 10 years, significant liver disease with AST and ALT more than 3 times the normal range.
6. Concomitant medications that will alter the pharmacodynamic/pharmacokinetic properties of the study medication. Participant who are taking the following medications: Amprenavir; Atazanavir; Clarithromycin; Delavirdine; Diclofenac; Fosamprenavir; Imatinib; Indinavir; Isoniazid; Itraconazole; Ketoconazole; Miconazole; Nefazodone; Nelfinavir; NiCARdipine; Propofol; Quinidine; Ritonavir; Telithromycin; Phenytoin; carbamazepine and phenobarbital
7. Subjects on psychoactive medications must be on a stable dose more than 3 months
8. Female subjects who are pregnant or nursing.
9. Subject is facing future imprisonment.
10. A known allergy to zonisamide or sulfa.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2006-11; Primary Completion 2007-10 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ofra Sarid-Segal, MD, Principal Investigator — Boston University
Locations (1):
- Boston University Medical Campus, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Zonisamide-Placebo Sessions: In this within subjects study, subjects received zonisamide in one session and placebo in a second
Period: Overall Study
Arm/Group | Zonisamide-Placebo Sessions
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Zonisamide-Placebo Sessions
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Grams Ethanol Consumed During Second Hour of the Alcohol Self-Administration Sessions
Description: Grams Ethanol Consumed During Second Hour of the Alcohol Self-Administration Sessions for Zonisamide and Placebo Conditions
Time Frame: 1 day
Population: This was a laboratory based study. An ITT analysis was used.
Measure: Mean (Standard Error); unit: Grams
Arm/Group | Zonisamide-Placebo Sessions
Number analyzed (Participants) | 10
Grams
  Zonisamide | 9.0 (3.7)
  Placebo | 18.2 (3.1)
Statistical Analysis 1: Comparison: Zonisamide-Placebo Sessions; The analysis involved a within subjects comparison. The null hypothesis was that there would be no difference in the amount of ethanol consumed in either the first or second hour of self-administration sessions. Results presented here are for the second hour of the self-administration sessions; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Results presented are for post-hoc comparisons of least squares means with Tukey-Kramer adjucted p values; Mean Difference (Final Values) = -9.2, Standard Error of Mean 3.4 — The estimated value is for the difference between the means obtained for the second hour of the self-administration sessions for the placebo and zonisamide conditions

2. Secondary Outcome: Score Digit Symbol Modalities Test
Description: Difference score between zonisamide and placebo treatment conditions for the Digit Symbol Modalities Test scores obtained 40 minutes after ingestion of a priming dose of ethanol.This test involves transcribing from a key in which numbers appear below a series of symbols to boxes below symbols matched to those in the key. This task must be completed in 90 nseconds. This test measures visuomotor speed and aspects of attention. Scoring is the total number of correctly transcribed numbers. The maximum score on this test 110 points.
Time Frame: 40 minutes post alcohol ingestion
Population: ITT
Measure: Mean (Standard Error); unit: Numeric Score
Arm/Group | Zonisamide-Placebo Sessions
Number analyzed (Participants) | 10
Numeric Score | 2.2 (5.7)
Statistical Analysis 1: Comparison: Zonisamide-Placebo Sessions; Null hypothesis: No difference in DSMT scores for zonisamide and placebo treatments 40 minutes after ingestion of ethanol; Test type: Superiority or Other; p = 0.61, Mixed Models Analysis — P value shown is for a post-hoc comparison of least squares means generated by the mixed model used; Mean Difference (Final Values) = 2.2, Standard Error of Mean 5.7 — Analysis for difference between DSMT scores at 40 minutes post alcohol ingestion for zonisamide and placebo involved post-hoc comparisons of least squares means

ADVERSE EVENTS:
Arm/Group | Zonisamide-Placebo Sessions
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes